CLINICAL TRIAL: NCT06825663
Title: Brain Insulin Resistance Index in Plasma Neuronal Exosomes As Predictive Biomarkers of Alzheimer's Disease
Brief Title: Marker of Brain Insulin Resistance in AD Prognosis
Acronym: IREN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Thérèse Jonveaux (Unknown); Laure Joly (Unknown)
Responsible Party: Principal Investigator, Catherine MALAPLATE, Dr, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A00609-38
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-05

CONDITIONS: Prognosis Biomarker of AD; Mild Cognitive Impairment; Brain Insuline Resistance
Keywords: Alzheimer' disease; biomarker; Blood neuronal exosomes; Brain insuline resistance
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MCI (Experimental): Men or women aged 18 to 75 followed for mild cognitive disorders at the Nancy CHRU CMRR for 1 to 2 years
  Interventions: Biological: Blood punction

INTERVENTIONS:
Biological: Blood punction — At each annual visit (+/- 3 months), 4X10 mL blood will be taken (1 dry tube, 1 heparinised tube, 2 EDTA tubes)

SUMMARY:
Basic research data from the literature on the links between cerebral insulin resistance and Alzheimer's disease (AD) suggest that this pathophysiological mechanism is involved at a very early stage in the development of the disease.

The insulin receptor (IR) is a tyrosine kinase receptor whose activation by insulin binding leads to autophosphorylation of its IRβ subunits and then of the insulin receptor substrate proteins (IRS-1). The ratio of IRS residues phosphorylated on serine 312 (P(Ser312)-IRS-1) to total phosphorylated IRS or IRS phosphorylated on its tyrosines has been proposed by some authors as an index of insulin resistance in the brain. IRS-1 proteins can be measured in exosomes, and in particular in neuronal exosomes isolated from plasma. It is therefore conceivable to measure this index in these biological samples specifically derived from neurons and available from a simple blood test, in order to determine whether it could be of prognostic interest in patients with mild cognitive impairment (MCI), in particular by making it possible to identify at an early stage patients who are going to convert to AD.

DETAILED DESCRIPTION:
Basic research data from the literature on the links between cerebral insulin resistance and AD suggest that this pathophysiological mechanism is involved at a very early stage in the development of the disease. The multiple effects of insulin on cerebral bioenergetic regulation, synaptic viability, dendritic spine formation and neurotransmitter turnover, as well as on the clearance and degradation of Aβ peptide, All these factors suggest that dysregulation of insulin signalling pathways in the brain may contribute early on to neurodegeneration in AD, and represent both a therapeutic lever and a source of biomarkers relevant to diagnosis and prognosis (1). Several clinical trials are currently underway to validate the value of insulin administration or the use of drugs that affect insulin receptor sensitivity in the treatment of AD patients (2).

Given these arguments in favour of the role of cerebral insulin resistance in the early stages of AD, being able to measure such an index in plasma could prove invaluable in the management of patients. However, it is still difficult to distinguish between peripheral and central origin of the molecules measured, which explains the frequent use of lumbar puncture to diagnose neurological diseases. An alternative strategy could be based on the specific isolation of neuronal exosomes present in the blood. Exosomes are vesicles derived from late endosomes and containing nucleic acids, proteins and lipids. Specific protein markers, such as L1CAM for neurons, enable them to be isolated by immunoaffinity, according to their cellular origin. It is then possible to measure plasma biomarkers whose neuronal origin is certain (4).

IRS-1 proteins can be measured in exosomes, and in particular in neuronal exosomes isolated from plasma, but studies on the use of this index in AD are rare. One team of researchers has taken a particular interest in this question, showing that the insulin resistance index is significantly higher in AD patients than in control subjects or those with another neurodegenerative disease (3). A more recent study also showed that, in Alzheimer's subjects, brain volume was positively correlated with the level of IRS-1 phosphorylated on its tyrosine residues, whereas it was negatively correlated with the level of IRS-1 phosphorylated on serine 312 (5). This index in exosomes has also been proposed to distinguish good from poor responders to insulin treatment (6) or to illustrate the links between amyloid and Tau pathologies in AD (7). To date, no study has proposed using this index in plasma neuronal exosomes as a marker of conversion to AD in patients with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 75
* Have been treated for mild cognitive impairment at the Nancy CHRU CMRR for 1 to 2 years
* Person affiliated to a social security scheme or beneficiary of such a scheme
* Person who has received full information on the organisation of the research and has signed an informed consent form

Exclusion Criteria:

* Adult subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* A person who has converted to clinically proven AD. The fact that an LP to measure AD markers has been performed is not a criterion for inclusion.
* An adult unable to give consent
* Person deprived of liberty by a judicial or administrative decision
* Persons under psychiatric care by virtue of articles L. 3212-1 and L. 3213-1.
* Pregnant women, women in labour or breastfeeding mothers
* Persons staying in a health or social establishment for purposes other than research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
prognostic performance of insulin resistance indexes | 3 years
  Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value of Pser312-IRS1/Ptyr-IRS1 and Pser312-IRS1/IRS1 ratios measured at t0 (inclusion visit) Threshold value for these ratios to predict conversion to AD to be defined (no thresholds for these ratios in the literature) Conversion to AD defined by the clinician according to usual practice

SECONDARY OUTCOMES:
prognostic performance of insulin resistance indexes in diabetic and non-diabetic MCI patients | 3 years
  Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value of Pser312-IRS1/Ptyr-IRS1 and Pser312-IRS1/IRS1 ratios measured at t0 (inclusion visit) Threshold value for these ratios to predict conversion to AD to be defined (no thresholds for these ratios in the literature) Conversion to AD defined by the clinician according to usual practice
Link between cerebral insulin resistance index and conversion time | 3 years
  Time between date of first symptoms and date of conversion to AD in months Value of Pser312-IRS1/Ptyr-IRS1 and Pser312-IRS1/IRS1 ratios measured at t0 (inclusion visit) Conversion to AD defined by the clinician according to usual practice
Link between cerebral insulin resistance index and glycated haemoglobin level | 3 years
  Pser312-IRS1/Ptyr-IRS1 and Pser312-IRS1/IRS1 ratios measured at t0 (inclusion visit) HbA1c in % measured at t0 (inclusion visit)
Link between cerebral insulin resistance index and vascular resistance | 3 years
  Pser312-IRS1/Ptyr-IRS1 and Pser312-IRS1/IRS1 ratios measured at t0 (inclusion visit) Vascular resistance measured at t0 (inclusion visit)